CLINICAL TRIAL: NCT00979758
Title: Strengthening Transplantation Effects of Bone Marrow Mononuclear Cells With Atorvastatin in Myocardial Infarction
Acronym: STEM-AMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yuejin Yang, Vice president of Fuwai hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Fuwai Hospital 2009
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Myocardial Infarction; Stem Cell Transplantation; Angioplasty, Transluminal, Percutaneous Coronary
MeSH Terms: conditions — Myocardial Infarction | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Atorvastatin (Sham Comparator): Atorvastatin routine dose
  Interventions: Drug: Atorvastatin and mononuclear cells transplantation
- Intensive Atorvastatin (Placebo Comparator): Atorvastatin Intensive dose
  Interventions: Drug: Atorvastatin and mononuclear cells transplantation
- Atorvastatin+Transplantation (Active Comparator): Atorvastatin routine dose+ Mononuclear cells Transplantation
  Interventions: Drug: Atorvastatin and mononuclear cells transplantation
- Intensive Atorvastatin+Transplantation (Experimental): Atorvastatin intensive dose+ Mononuclear cells Transplantation
  Interventions: Drug: Atorvastatin and mononuclear cells transplantation

INTERVENTIONS:
Drug: Atorvastatin and mononuclear cells transplantation — Routine or intensive dose of Atorvastatin therapy and mononuclear cells transplantation
  Other Names: Statin; Bone marrow stem cells transplantation

SUMMARY:
The benefit of current stem cell transplantation therapy for myocardial infarction is limited by low survival rate for stem cell. The purpose of this study is to test whether intensive Atorvastatin therapy can improve the outcome of patients with impaired left ventricle function after myocardial infarction who underwent intracoronary transfer of autologous bone marrow cells.

DETAILED DESCRIPTION:
The major challenge to a successful stem cell therapy for myocardial infarction is the low survival rate of implanted cells in the damaged tissue. Atorvastatin, an HMG-CoA reductase inhibitor, has multiple biological activities independent of cholesterol-lowering action.This study is performed to find out more information about the strategy with Atorvastatin therapy to improve the survival of implanted cells. autologous bone marrow stem cells transplantation. Patients between 30 and 80 years of age who receive autologous bone marrow stem cell transplant at the Fuwai cardiovascular hospital may be eligible for this study. These patients receive autologous bone marrow cells transplantation intracoronary undergoing Percutaneous Coronary Intervention with regular or high dose of Atorvastatin treatment. The objective evaluations will be performed at baseline and during 12 months follow-up.

Heart function tests may include the following:

1. Electrocardiogram (EKG) evaluates the electrical activity of the heart. Electrodes placed on the chest transmit information from the heart to a machine.
2. Echocardiogram (Echo) is an ultrasound test that uses sound waves to create an image of the heart and examine the function of the heart chambers and valves.
3. Gated acquisition scan is a nuclear medicine test that uses a small amount of radioactive chemical injected into a vein. A special scanner creates an image of the heart for examining the beating motion of the muscle.
4. MRI evaluates function of the heart chambers the beating motion of the muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with coronary disease undergoing PCI.
2. At most 2 months since last episode of ST-elevation myocardial infarction.
3. Left ventricular ejection fraction >=20% <=45% based on coronary angiography or echocardiography.

Exclusion Criteria:

Any one of the following exclusion criteria is sufficient to disqualify a patient from the study.

1. Patients with non-ST-elevation myocardial infarction.
2. Patients with normal left ventricular function.
3. Patients with mechanical complications of myocardial infarction.
4. Patients with a malignant tumor.
5. Patients with infection disease.
6. Less than 6 months since last episode of stroke.
7. Patients with hematological disease (leukemia, myeloproliferative disease, or myelodysplastic syndromes).
8. AST (GOT) exceeding 100 IU/L or ALT (GPT) exceeding 100 IU/L.
9. Leukocytes less than 4,000/µL or exceeding 10,000/µL.
10. Platelets less than 100,000/µL.
11. Hemoglobin less than 10 g/dL.
12. Pregnant or nursing patients, those who may be pregnant, or those who plan on becoming pregnant before the end of the study period.
13. Any other reason that the Clinical Supervisors or Clinical Researchers may have for considering a case unsuitable for the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in left ventricular ejection fraction from baseline to 12 months' follow-up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yang yuejin, Doctor, Study Director — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, China

REFERENCES:
- [Derived] Yang YJ, Qian HY, Song L, Geng YJ, Gao RL, Li N, Wang H, Tian XQ, Huang J, Huang PS, Xu J, Shen R, Lu MJ, Zhao SH, Wu WC, Wu Y, Zhang J, Qian J, Xu JY, Xiong YY. Strengthening effects of bone marrow mononuclear cells with intensive atorvastatin in acute myocardial infarction. Open Heart. 2020 May;7(1):e001139. doi: 10.1136/openhrt-2019-001139. PMID 32393654